CLINICAL TRIAL: NCT00916604
Title: A Randomized, Single-blind, Placebo-Controlled, Multi-centre, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Multiple Ascending Oral Doses of AZD1656 in Japanese T2DM Patients
Brief Title: To Study Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD1656 in Japanese Type 2 Diabetes Mellitus (T2DM) Patients
Acronym: JMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof, Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1020C00004
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Type 2 Diabetes
Keywords: AZD1656; Safety; Pharmacokinetics; Pharmacodynamic; Multiple ascending doses; Japanese; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- A (Experimental): 3 gradually increasing repeated oral doses of AZD1656 given to 3 groups (6 on active substance in each group)
  Interventions: Drug: AZD1656
- B (Placebo Comparator): Placebo oral suspension given to 3 groups (2 on placebo in each group)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — Three increasing dose-steps with oral suspension, 8 days treatment
  Arms: A
Drug: Placebo — Placebo oral suspension, 8 days treatment
  Arms: B

SUMMARY:
The purpose of this study is to assess the safety and tolerability of AZD1656 after multiple repeated oral doses in Japanese patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female non-childbearing potential Japanese T2DM patients, 30-75 years.
* A body mass index (BMI) of 19 to 27 kg/m2.
* Diagnosed Diabetes Mellitus patients treated with diet and exercise or with up to two oral anti-diabetic drugs. Stable glycemic control indicated by no changed treatment within 3 months prior to enrollment.

Exclusion Criteria:

* Renal dysfunction GFR < 60 mL/min.
* Systolic pressure (SBP) > 160 mmHg or diastolic pressure (DBP) > 95 mmHg
* Clinically significant illness or clinically relevant trauma, as judged by the investigator, within two weeks before the first administration of the IP.
* History of ischemic heart disease, stroke, transient ischemic attack or symptomatic peripheral vascular disease.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-05; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety by assessment of adverse events, BP, pulse rate, plasma glucose, safety laboratory variables and ECG | Blood samples taken repeatedly during 24 hours on study day sessions

SECONDARY OUTCOMES:
Pharmacokinetic variables (AUC, Cmax, tmax, t½, CL/F, Ae and CLR). | Blood samples taken repeatedly during 24 hours on study day sessions
Pharmacodynamic variables (P-Glucose, S-Insulin and S-C-peptide). | Blood samples taken repeatedly during 24 hours on study day sessions

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, Study Director — AstraZeneca R&D Mölndal; Takashi Eto, MD, PhD, Principal Investigator — PS Clinic, Fukuoka, Japan; Mitsuyasu Hokamura, MD, Principal Investigator — HONJO CLINIC II, Tokyo, Japan
Locations (2):
- Japan (2):
  - Research Site, Fukuoka
  - Research Site, Tokyo